CLINICAL TRIAL: NCT01532596
Title: The Effects of Mindfulness Meditation in Older Adults
Brief Title: Mindfulness Meditation in Older Adults
Acronym: MIND
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, J. David Creswell, Post-Doctoral Fellow, Cousins Center for Psychoneuroimmunology, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MBSR-Older-00001
Record Dates: First submitted 2012-02-08; First posted 2012-02-14 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Aging
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): A standardized 8-week mindfulness meditation training program
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Wait-List (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — 8-week standardized mindfulness meditation training program
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction

SUMMARY:
The purpose of this study is to test if an 8-week mindfulness meditation training (vs a wait-list control condition) program reduces neurobehavioral reactivity and improves affect regulation in a sample of older adults, as measured by functional magnetic resonance imaging. Additionally, we will examine if mindfulness meditation training reduces loneliness and markers of chronic inflammation.

DETAILED DESCRIPTION:
It is well established that mindfulness meditation interventions improve a wide-range of mental and physical health outcomes in stressed patient populations, although the underlying mechanisms are currently unknown. It has been suggested that mindfulness training may reduce reactivity to stimuli and improve regulation, although these mechanisms have not been examined (using functional neuroimaging). Additionally, it is well-established that loneliness and inflammation are major risk factors for morbidity and mortality in older adults, although it is currently unknown whether mindfulness meditation training may reduce these risk factors. The purpose of the proposed study is to test if mindfulness meditation training (vs a wait-list control condition) reduces neurobehavioral reactivity and improves affect regulation in a sample of healthy older adults, as measured by functional magnetic resonance imaging. Additionally, we will examine whether mindfulness meditation training reduces loneliness and markers of inflammation.

Participants will be recruited in the Los Angeles area and randomly assigned to the 8-week Mindfulness-Based Stress Reduction (MBSR) intervention or to a wait-list. All participants will provide a blood sample and complete a psychosocial survey before and after the intervention, and complete a 60-minute neuroimaging assessment before and after the MBSR program. All participants who are randomly assigned to the wait-list will be offered the MBSR intervention after the 8-week intervention period and then complete an additional post-test assessment after completing the MBSR program (which will include a blood sample, psychosocial survey, and a neuroimaging assessment). Participants will complete neuroimaging tasks (where they will be presented with words, pictures, and sounds) before and after receiving the MBSR intervention, which will assess neural activity and regulation responses before and after mindfulness meditation training.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults between the ages of 55-85 years of age at time of entry
* post-menopausal and not pregnant (women only)
* Accessible geographically and willing to come to UCLA for all study related activities

Exclusion Criteria:

* they have regularly (>1 time per week) practiced a mind-body therapy anytime in the last six months (e.g., meditation, yoga, tai chi)
* are not ambulatory, (c) indicate any treatment for mental health problems in the last six months
* indicate any major physical health problems in the last three months
* use medications affecting cardiovascular or endocrine function
* are left-handed
* or have metal in their bodies (including pacemakers and permanent piercings (e.g., bellyrings), but not dental fillings)
* indicate regular use of psychotropic medication or psychotherapy in the last six months
* cognitive impairment as indicated by a score lower than 23 on the Mini-Mental State examination
* smokers
* indicate feeling claustrophobic in confined spaces, such as an fMRI scanner
* weigh over 300 lbs
* indicate any use of doctor prescribed cholesterol lowering medications (e.g., statins)
* use any doctor prescribed pain medication
* indicate any implants

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Functional Neural Activity | Change from Baseline to 2 months
  Neural responses to emotionally evocative stimuli

SECONDARY OUTCOMES:
Pro-inflammation | Change from Baseline to 2 months
  Genetic and protein measures of inflammation
Loneliness | Change from Baseline to 2 months
  self-reported loneliness
Psychological Distress | Change from Baseline to 2 months
  self-reported psychological distress

CONTACTS AND LOCATIONS:
Overall Officials: J. David Creswell, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Cousins Center for Psychoneuroimmunology, UCLA, Los Angeles, California, United States